CLINICAL TRIAL: NCT06149975
Title: Feasibility of a Motor-cognitive Training Program in Patients With Traumatic Brain Injury During Acute Hospitalization
Brief Title: Feasibility of a Motor-cognitive Training Program in Patients With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Eleftheria Giannouli, Principal Investigator, Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: StepIt TBI
Record Dates: First submitted 2023-10-22; First posted 2023-11-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Traumatic Brain Injury
Keywords: motor-cognitive training; dual-task; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): In addition to the usual care, the study participants receive the motor-cognitive training "StepIt". The "StepIt" will be conducted as an approximately 15-minute one on one training for at least 3 to max. 10 sessions during the stay at the hospital.
  Interventions: Other: motor-cognitive training

INTERVENTIONS:
Other: motor-cognitive training — The motor-cognitive training in this study will be conducted in form of a step-based dual-task training. A mat (approximately 90 x 90 cm) made from extra non-slip yoga mats is required. The mat is divided into 9 equal squares with a 3 x 3 pattern. Participants will be presented with stepping patterns which they must memorize and then execute on the mat in the pace given by a metronome. All participants will start at the same level. The progression will be adjusted individually according to the fixed criteria of the "StepIt" concept within the sessions. All sessions will be supervised by at least one physical therapist.

SUMMARY:
The goal of this clinical study is to test feasibility of a motor-cognitive training program in patients after mild to severe traumatic brain injury in an acute hospitalization setting.

The intervention is a step-based dual-task training, i.e. patients are presented with step patterns that they have to memorize and then execute in the tempo given by a metronome.

Researchers will assess the feasibility of the motor-cognitive training regarding acceptance and safety, user evaluation of the training and training performance.

DETAILED DESCRIPTION:
A traumatic brain injury (TBI) refers to a functional disorder of the brain with or without demonstrable injuries to the brain as a result of external force to the skull and/or brain. The most common causes are traffic accidents and falls. After TBI, impairments may occur in motor skills such as gait stability, static and dynamic balance and motor coordination as well as cognitive skills such as memory, dual- and multi-tasking (DT/MT), and psychomotor speed. Therefore, rapid improvement of motor and cognitive functioning and falls prevention are essential.

Dual-task training have been shown to improve gait performance and to reduce the risk of falling in some neurological disorders, such as Parkinson's disease and stroke. Although there are differences in the underlying pathophysiology between these neurological conditions and TBI, research has identified many common fall-risk factors and thus it can be expected that TBI patients would also profit from cognitive-motor dual-task training. However, research on the effects of such training in TBI patients in scarce. To our knowledge, there is only one study that has looked into the effects of dual-task motor-cognitive training in people with neurological conditions, including (but not specifically for) persons with TBI. For this reason, this study aims to assess the feasibility of a concept for stepping training (StepIt) that addresses motor as well as cognitive falls-related aspects in patients with TBI.

This study will be conducted as one-arm, monocentric intervention trial. After admission to the normal ward, patients potentially fulfilling the eligibility criteria will be informed orally and in writing about the study and asked if they wish to participate. All interested participants will then be screened for final inclusion. Baseline data collection will occur prior to the first training session and training evaluation will be conducted after 3 to max. 10 trainings (depending on the length of their hospital stay). During each training session individual training parameters will be documented. In addition to the usual care, the study participants receive the motor-cognitive training "StepIt". The "StepIt" will be conducted as an approximately 15-minute one on one training for at least 3 to max. 10 sessions during the stay at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with mild (Glasgow Coma Scale 14-15), moderate (Glasgow Coma Scale 9-13) or severe (Glasgow Coma Scale 3-8) TBI
* Age ≥ 18 years
* Planned hospital treatment >24h on regular ward (non-ICU)
* Physically able to stand (using cane if needed)
* Able to give informed consent

Exclusion Criteria:

* Limited vision and hearing ability (except facial injuries with monocular swelling)
* Inability or contraindications to undergo the investigated intervention.
* ICU stay only
* Montreal Cognitive Assessment (MoCa) score < 16

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | through study completion, an average of 9 months
  Number of patients fitting to the inclusion exclusion (resp. exclusion) criteria as percentages of persons with TBI admitted in the hospital during the study period
Inclusion rate | through study completion, an average of 9 months
  Number of patients included in the study as percentages of patients fitting to the inclusion (resp. exclusion) criteria
Attrition rate | through study completion, an average of 9 months
  Number of Drop-outs as percentages of patients included in the study
Adherence rate | through study completion, an average of 9 months (over all training sessions)
  Number of attended training sessions as percentages of total possible training sessions
Compliance rate | through study completion, an average of 9 months (over all training sessions)
  Number of attended training minutes as percentages of the total possible training minutes
Security incidents | through study completion, an average of 9 months (over all training sessions)
  Total number of (Serious) Adverse Events (SAE/AE)

SECONDARY OUTCOMES:
Physical and cognitive load | through study completion, an average of 9 months (after each training session (min. 3 times max. 10 times))
  Physical and cognitive load assessed with the National Aeronautics and Space Administration-Task Load Index (NASA-TLX). The NASA-TLX is a self-report, multidimensional assessment tool that rates perceived workload in order to assess a task, a system, or other aspects of performance (in this case the "StepIi" trainings). It contains five subscales: Mental Demand, Physical Demand, Temporal Demand, Performance, Effort and Frustration. Each subscale can be given a score between 0 and 20. A higher score reflects a higher workload.
Patient Satisfaction | through study completion, an average of 9 months (after each training session (min. 3 times max. 10 times))
  With a tailored (self-made) usability questionnaire the patient satisfaction will be assessed. The questionnaire records how the participants felt about the training, how satisfied they were with the training and whether they would recommend the training to others. The questionnaire contains 13 questions (Yes-No questions, Likert-Scale, and open questions). Each item will be evaluated separately.
Improvement | through study completion, an average of 9 months (after each training session (min. 3 times max. 10 times))
  Comparison of the entry level versus the highest achieved level in percentage (for following training parameters: i. length of stepping sequence, ii.beats/minute, iii. Stepping sequence complexity)
Training capacity | through study completion, an average of 9 months (after each training session (min. 3 times max. 10 times))
  Number of taught patterns per training session

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Katrin Hickmann, PD Dr., Study Director — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital of St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Menon DK, Schwab K, Wright DW, Maas AI; Demographics and Clinical Assessment Working Group of the International and Interagency Initiative toward Common Data Elements for Research on Traumatic Brain Injury and Psychological Health. Position statement: definition of traumatic brain injury. Arch Phys Med Rehabil. 2010 Nov;91(11):1637-40. doi: 10.1016/j.apmr.2010.05.017. PMID 21044706
- [Background] Brazinova A, Rehorcikova V, Taylor MS, Buckova V, Majdan M, Psota M, Peeters W, Feigin V, Theadom A, Holkovic L, Synnot A. Epidemiology of Traumatic Brain Injury in Europe: A Living Systematic Review. J Neurotrauma. 2021 May 15;38(10):1411-1440. doi: 10.1089/neu.2015.4126. Epub 2018 Dec 19. PMID 26537996
- [Background] Galea OA, Cottrell MA, Treleaven JM, O'Leary SP. Sensorimotor and Physiological Indicators of Impairment in Mild Traumatic Brain Injury: A Meta-Analysis. Neurorehabil Neural Repair. 2018 Feb;32(2):115-128. doi: 10.1177/1545968318760728. PMID 29554850
- [Background] Rabinowitz AR, Levin HS. Cognitive sequelae of traumatic brain injury. Psychiatr Clin North Am. 2014 Mar;37(1):1-11. doi: 10.1016/j.psc.2013.11.004. Epub 2014 Jan 14. PMID 24529420
- [Background] Berkner J, Meehan WP 3rd, Master CL, Howell DR. Gait and Quiet-Stance Performance Among Adolescents After Concussion-Symptom Resolution. J Athl Train. 2017 Dec;52(12):1089-1095. doi: 10.4085/1062-6050-52.11.23. Epub 2017 Nov 20. PMID 29154694
- [Background] Spano B, De Tollis M, Taglieri S, Manzo A, Ricci C, Lombardi MG, Polidori L, Griffini IA, Aloisi M, Vinicola V, Formisano R, Caltagirone C, Annicchiarico R. The Effect of Dual-Task Motor-Cognitive Training in Adults with Neurological Diseases Who Are at Risk of Falling. Brain Sci. 2022 Sep 7;12(9):1207. doi: 10.3390/brainsci12091207. PMID 36138943
- [Background] Giannouli E, Morat T, Zijlstra W. A Novel Square-Stepping Exercise Program for Older Adults (StepIt): Rationale and Implications for Falls Prevention. Front Med (Lausanne). 2020 Jan 14;6:318. doi: 10.3389/fmed.2019.00318. eCollection 2019. PMID 31993435
- [Background] Fritz NE, Basso DM. Dual-task training for balance and mobility in a person with severe traumatic brain injury: a case study. J Neurol Phys Ther. 2013 Mar;37(1):37-43. doi: 10.1097/NPT.0b013e318282a20d. PMID 23364169
- [Background] Zhou Q, Yang H, Zhou Q, Pan H. Effects of cognitive motor dual-task training on stroke patients: A RCT-based meta-analysis. J Clin Neurosci. 2021 Oct;92:175-182. doi: 10.1016/j.jocn.2021.08.009. Epub 2021 Aug 25. PMID 34509248
- [Background] Silva RDN, Afonso SV, Felipe LR, Oliveira RA, Patrizzi Martins LJ, Pascucci Sande de Souza LA. Dual-task intervention based on trail making test: Effects on Parkinson's disease. J Bodyw Mov Ther. 2021 Jul;27:628-633. doi: 10.1016/j.jbmt.2021.04.013. Epub 2021 May 4. PMID 34391298
- [Background] Yang YR, Chen YC, Lee CS, Cheng SJ, Wang RY. Dual-task-related gait changes in individuals with stroke. Gait Posture. 2007 Feb;25(2):185-90. doi: 10.1016/j.gaitpost.2006.03.007. Epub 2006 May 2. PMID 16650766
- [Background] Liu YC, Yang YR, Tsai YA, Wang RY. Cognitive and motor dual task gait training improve dual task gait performance after stroke - A randomized controlled pilot trial. Sci Rep. 2017 Jun 22;7(1):4070. doi: 10.1038/s41598-017-04165-y. PMID 28642466
- [Background] Spano B, Lombardi MG, De Tollis M, Szczepanska MA, Ricci C, Manzo A, Giuli S, Polidori L, Griffini IA, Adriano F, Caltagirone C, Annicchiarico R. Effect of Dual-Task Motor-Cognitive Training in Preventing Falls in Vulnerable Elderly Cerebrovascular Patients: A Pilot Study. Brain Sci. 2022 Jan 27;12(2):168. doi: 10.3390/brainsci12020168. PMID 35203932
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223